CLINICAL TRIAL: NCT07086066
Title: Investigation of the Effectiveness of Diaphragm Mobilization on Range of Motion, Function, and Pain in Patients With Rotator Cuff Lesions
Brief Title: Diaphragm Mobilization With Rotator Cuff Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Muhammed Fatih Kavak, Dr. Physiotherapist, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61351342/020-827
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Rotator Cuff Syndrome
Keywords: pain; range of motion; function
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: There were two groups in the study. The experimental group received conventional physical therapy combined with diaphragm mobilization. The control group received only conventional physical therapy without diaphragm mobilization.
Who Masked: Participant
Masking Description: The participants were unaware of which group they had been assigned to. Based on the order of their arrival at the hospital, those who arrived first, third, fifth, and so on were assigned to the diaphragm mobilization group, while those who arrived second, fourth, sixth, and so on were assigned to the standard physiotherapy group. This allocation method ensured that participants remained blinded to their group assignment, minimizing potential bias in their responses or expectations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragm mobilization group (Experimental): The experimental group received conventional physical therapy and diaphragm mobilization.
  Interventions: Other: Diaphragm mobilization; Other: conventional physical therapy
- standard physiotherapy group (Active Comparator): The control group will receive only conventional physical therapy.
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: Diaphragm mobilization — This group underwent treatment three times a week, with each session lasting 40 to 60 minutes, over a period of six weeks. Diaphragm mobilization included techniques aimed at increasing muscle elasticity, improving postural balance, and reducing pain by stimulating the sympathetic and parasympathetic nervous systems. In each session, participants received 20 minutes of TENS and 10 minutes of cryotherapy. Following this, diaphragm mobilization was applied. During the application, participants were positioned comfortably in the supine position. The physiotherapist palpated the diaphragm, instructed the participant in diaphragmatic breathing, and asked them to take a deep diaphragmatic breath. During expiration, the diaphragm was mobilized in the posterior and inferior directions. This mobilization was performed 10 times per session. Following that, posterior glide and inferior glide techniques were performed.
  Arms: Diaphragm mobilization group
Other: conventional physical therapy — As with the experimental group, therapy will be delivered three times per week for six weeks, with each session lasting between 40 and 60 minutes. Each session will include 20 minutes of TENS and 10 minutes of cryotherapy, followed by posterior and inferior gliding techniques on the glenohumeral joint and capsular stretching. Functional exercises will also include wand exercises (two sets of 10 repetitions) and finger ladder exercises targeting shoulder flexion and abduction, but without the addition of diaphragm mobilization techniques.

SUMMARY:
The glenohumeral joint is the least restricted joint in terms of mobility compared to other joints in the human body. The rotator cuff is a part of the shoulder complex consisting of four muscles and their tendons, which are responsible for stabilizing the shoulder joint. These muscles are the supraspinatus, infraspinatus, teres minor, and subscapularis. The supraspinatus muscle enables shoulder abduction, infraspinatus and teres minor provide external rotation, and the subscapularis is responsible for internal rotation.

The presence of a rotator cuff lesion is the most common cause of shoulder pain. It usually results from the tear, inflammation, or injury of one or more rotator cuff muscles. It is more prevalent in elderly individuals and is characterized by severe shoulder pain, limited range of motion, and functional loss. These symptoms negatively impact the patient's performance and significantly reduce their quality of life.

The diaphragm is a large, dome-shaped muscle and the primary muscle of respiration. It is innervated by the phrenic nerve, which is connected to the vagus nerve. During breathing, the diaphragm's movements can directly or indirectly influence the sympathetic and parasympathetic nervous systems, thereby modulating pain perception in the body.

Moreover, there is a significant relationship between the shoulder and diaphragm in terms of myofascial connections and neural innervation. Effective functioning of the diaphragm not only contributes to proper respiration but also positively affects spinal mobility and overall posture. It supports the efficiency of upper body structures such as the cervical spine, shoulder, and neck.

Proper diaphragmatic function contributes to core stability, which in turn may reduce the load on shoulder structures. Manual techniques targeting the diaphragm can enhance its function, potentially reducing the mechanical load on the shoulder complex, alleviating pain, and improving the patient's overall functional capacity.

DETAILED DESCRIPTION:
This randomized controlled study aims to evaluate the clinical effects of diaphragm mobilization on joint range of motion, pain, and functional status in individuals diagnosed with rotator cuff lesions. The study will be conducted at Sancak Medical Physical Therapy Center between February 10, 2025, and March 15, 2025. Fifty volunteer participants, both male and female, aged between 25 and 55, will be included. All participants will have clinically diagnosed and radiologically confirmed rotator cuff injuries, accompanied by significant pain or functional limitation, indicated by a Visual Analog Scale (VAS) score greater than 3. Before participating in the study, each individual will provide informed consent.

Participants will be randomly assigned to one of two groups: the experimental group or the control group. Demographic information such as age, gender, occupation, educational status, and body mass index will be collected prior to treatment. Pain levels will be assessed using the Visual Analog Scale (VAS), a simple and widely accepted tool where 0 indicates no pain and 10 represents the most severe pain imaginable. Range of motion will be measured using a universal goniometer, specifically focusing on shoulder flexion, abduction, internal rotation, and external rotation angles. Functional capacity will be evaluated with the Upper Extremity Functional Index (UEFI), a self-reported questionnaire used to measure disability in individuals with upper extremity musculoskeletal disorders. The UEFI consists of 20 items, and the total score ranges from 0 to 80, with higher scores indicating better function.

Assessments will be carried out at baseline and repeated at the end of the six-week intervention period. The experimental group will receive a combination of conventional physical therapy and diaphragm mobilization. Treatment will occur three times per week, with each session lasting between 40 and 60 minutes over six consecutive weeks. Each session will begin with a 20-minute application of transcutaneous electrical nerve stimulation (TENS), followed by 10 minutes of cryotherapy. Diaphragm mobilization will then be performed while the participant lies in a relaxed supine position. The physiotherapist will palpate the diaphragm and teach the participant diaphragmatic breathing techniques. During expiration, the diaphragm will be mobilized in a posterior and inferior direction. This process will be repeated 10 times in each session. Following diaphragm mobilization, the therapist will apply posterior and inferior gliding techniques to the glenohumeral joint, followed by capsular stretching. Functional rehabilitation will include wand exercises performed in two sets of 10 repetitions and finger ladder exercises involving shoulder flexion and abduction.

The control group will receive only conventional physical therapy. As with the experimental group, therapy will be delivered three times per week for six weeks, with each session lasting between 40 and 60 minutes. Each session will include 20 minutes of TENS and 10 minutes of cryotherapy, followed by posterior and inferior gliding techniques on the glenohumeral joint and capsular stretching. Functional exercises will also include wand exercises (two sets of 10 repetitions) and finger ladder exercises targeting shoulder flexion and abduction, but without the addition of diaphragm mobilization techniques.

This study is designed to investigate whether incorporating diaphragm mobilization into a traditional rehabilitation program yields superior outcomes in reducing pain, improving joint mobility, and enhancing upper extremity function compared to conventional therapy alone. By examining the neuromuscular and postural influences of the diaphragm, the study seeks to identify a potentially valuable and underutilized therapeutic technique that could support shoulder rehabilitation protocols, particularly in individuals with rotator cuff pathology.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged between 25 and 55

Individuals diagnosed with a rotator cuff injury through radiological methods

Individuals experiencing severe pain (VAS ≥ 3) and functional loss

Individuals who are willing to participate in the study and have signed the written informed consent form after understanding the purpose and procedure of the study

Exclusion Criteria:

Individuals with a history of rotator cuff surgery

Individuals with a history of shoulder subluxation

Individuals with a history of SLAP lesions

Individuals with respiratory system diseases

Individuals with nerve damage (e.g., brachial plexus lesions) or neurological disorders that may affect shoulder movements

Individuals with psychological disorders (e.g., depression, anxiety) that may affect pain perception

Pregnant or breastfeeding women

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
range of motion | through study completion, an average of 3 months
  The range of motion will be evaluated using a universal goniometer to measure and document the angles of shoulder flexion, abduction, internal rotation, and external rotation. This instrument allows for reliable and standardized joint angle assessments, contributing to accurate monitoring of mobility improvements throughout the intervention.
subjective pain | through study completion, an average of 3 months.
  The Visual Analog Scale (VAS) will evaluate heel pain by asking participants to mark their pain level on a 10 cm scale, where 0 means no pain and 10 signifies severe pain, based on their experience over the past week.
Upper extremity function | through study completion, an average of 3 months
  The "Upper Extremity Functional Index" will be used for functional assessment. The Upper Extremity Functional Index is a self-administered questionnaire that measures disability in individuals with upper extremity orthopedic conditions. The questionnaire includes 20 activities, and the patient is asked to rate the difficulty of completing each activity. The scores from the 20 questions are summed to obtain a maximum possible score of 80. The lowest possible score is 0. Lower scores indicate greater difficulty in performing upper extremity activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)